CLINICAL TRIAL: NCT03023137
Title: Walking and Dietary Modification for Women With Consecutive Early Miscarriages: a Randomized Study
Brief Title: Walking and Dietary Modification for Recurrent Early Miscarriages
Acronym: W&D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital dos Servidores do Estado do Rio de Janeiro (Other Government)
Responsible Party: Principal Investigator, Silvia Hoirisch Clapauch, Principal Investigator, Hospital dos Servidores do Estado do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HospitalSERJ
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Recurrent Miscarriage
Keywords: prevention; carbohydrate; exercise; neonatal hypoglycemia
MeSH Terms: conditions — Abortion, Habitual; Motor Activity | interventions — Walking; Diet Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants were not blinded, but visits of the two groups were scheduled so as to not coincide..
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walking & dietary modification (W&D) (Active Comparator): W&D should begin when participants wish to conceive. The intervention was standardized by training of research staff. Careful instructions about walking speed and diet would be given to participants assigned to W&D at enrolment and at each consultation.
  Interventions: Behavioral: Walking & dietary modification
- Controls (No Intervention): No recommendations regarding diet or physical activity were given to controls. Antiemetics such as ondansetron would be given to controls complaining of vomiting.

INTERVENTIONS:
Behavioral: Walking & dietary modification — 1. Daily walking at a moderate pace (4 km/h) > 40 min, 7/7. Those remaining seated most of the day should walk 25-30 min twice a day, avoiding >12 h of physical inactivity. Walking may be replaced by stationary bicycle rides or swimming when convenient, which often occurred near term and when the mother was obese.
  2. At least two daily servings of protein-rich food (≥ 4 g/kg of meat, poultry, fish or eggs) per day. Avoidance of high-carbohydrate, low-fiber meals, such as snacks, candies, fiber-free juices, coconut water or sugar-sweetened beverages. Sucralose could be used as a sweetener. Participants are recommended to use ondansetron for nausea and vomiting prevention
  Other Names: W&D
  Arms: Walking & dietary modification (W&D)

SUMMARY:
This study is part of a big one aiming to evaluate how lifestyle interventions during pregnancy affect obstetric results, neonatal metabolism and the intelligence of the offspring (study not yet completed). Data regarding obstetric and neonatal results were entered in NCT01409382, but we decided to split results in two for the sake of clarity.

A cohort of women with early pregnancy losses without antiphospholipid antibodies was selected for two reasons. One is that these women follow strictly the recommendadtions. The second is that no medication has been shown to increase the rate of take-home babies in women with early miscarriages who test negative for antiphospholipid antibodies. We decided to focus on the fibrinolytic system because trophoblast migration and placental vasculogenesis and angiogenesis depend on plasmin-dependent extracellular matrix remodeling. Plasminogen activator inhibitor (PAI)-1 inhibits the generation of plasmin. Since both glucose and insulin increase PAI-1 synthesis, hyperglycemia itself, or by stimulating insulin production, reduces plasmin generation, which may impair placentation.

Abnormalities in glucose metabolism may be also deleterious to embryos by causing epigenetic changes. Chromosomal abnormalities are considered an important cause of early pregnancy losses.

Several lines of evidence lend support to the hypothesis that carbohydrate metabolism abnormalities contribute to the pathogenesis of recurrent early pregnancy losses. One is that of the pregnancies of the women with polycystic ovary syndrome, around 30 and 50% end with first-trimester miscarriages. Hyperinsulinemia is a prevalent feature of the syndrome, and interventions proven effective in reducing insulin levels, such as metformin, have been shown to reduce the rate of early miscarriages. The other is that patients with body mass index of ≥25 kg/m2 have significantly higher odds of early miscarriage, regardless of the method of conception.

The investigator's hypothesis was that a balanced diet combined to regular exercise, by improving glucose homeostasis, would increase the take-home baby rate in women with consecutive early miscarriages. Moderate exercises are usually well tolerated not only by the mother, but also by the fetus, as indicated by tests of fetal well-being, including umbilical artery systolic to diastolic ratio.

DETAILED DESCRIPTION:
Women aged 18 to 40 years trying to conceive spontaneously were eligible if they had two or more consecutive pregnancy losses in the first trimester, documented by pathology or ultrasound-confirmed gestational sac.

All participants underwent ultrasound examination before inclusion in the study. Exclusion criteria were any of the following: anatomic anomalies that may increase the risk of pregnancy losses, not amenable to surgical correction during pregnancy, such as uterine septum; antiphospholipid antibodies; prior second- or third-trimester losses; current multiple gestation; disabilities such as hemiplegia or paraplegia; renal or liver failure; conditions requiring a priori anticoagulation.

Participants were enrolled by staff at the participating center. Randomization to the intervention protocol Walking and Diet (W&D) or to a control group was performed before pregnancy occurred by a statistician using a computer-generated random-number table. This was not a double blind study, but care was taken to ensure that appointments of the patients assigned to the intervention protocol did not coincide with those of controls.

The intervention was standardized by training of research staff. Women assigned to W&D were instructed to walk at a moderate pace (4 km/h) for at least 40 minutes, seven days a week. Besides, those who remained seated most of the day were advised to walk 25 to 30 minutes twice a day, avoiding hence more than 12 hours of physical inactivity. Walking could be replaced by stationary bicycle rides or swimming when convenient, which often occurred near term and when the mother was obese. Strenuous exercises were discouraged.

Patients assigned to protocol W&D were also informed of the importance of a balanced diet and recommended to avoid high-glycemic index meals (high-carbohydrate, low-fiber). Sucralose could be used as a sweetener. As a strategy to promote satiety and reduce carbohydrate intake, W&D participants were also advised to eat at least two daily servings of protein-rich food. The intervention began when participants wished to conceive, continuing until delivery. Careful instructions about walking speed and diet were given to participants assigned to W&D at enrolment and at each consultation. During exercise, neither fetal nor maternal cardiac rate were assessed.

Non-adherence to the intervention protocol was suspected when non-obese participants assigned to W&D gained > 1 kg in 4 weeks until the 28th week of gestation, > 1.5 kg from the 28th to the 32nd week, and > 2 kg in 4 weeks thereafter, in the absence of edema. The threshold was lower for obese participants: > 700 g in 4 weeks until the 28th week of gestation, > 1 kg from the 28th to the 32nd week, and > 1.5 kg in 4 weeks thereafter21. Excessive weight gain aroused the suspicion of protocol violation because high carbohydrate consumption, especially when combined with physical inactivity stimulates the pancreas to overproduce insulin, a hormone that promotes fat storage. To enhance adherence to the protocol, W&D participants who gained excessive weight were recommended to increase the frequency, duration and intensity of the physical activity and to increase the protein intake. Participants of the W&D group who had a successful pregnancy volunteered to encourage mothers assigned to the intervention protocol, especially those who gained excessive weight.

At enrollment and during first-trimester consultations, W&D participants were explained that antiemetics such as ondansetron should be taken before nausea became severe, in order to help them tolerate balanced meals.

No recommendations regarding diet or physical activity were given to controls. Antiemetics such as ondansetron were given to controls who complained of hyperemesis.

All participants were given folic acid tablets 5 mg daily until 14 weeks of gestation, as prevention of neural tube defects. In both groups, participants reporting abdominal pain, cramps, and vaginal bleeding during the first-trimester were medicated with vaginal progesterone. Subcutaneous heparin was given to all participants whose pregnancies were complicated with nephrotic range proteinuria or any evidence of placental insufficiency. Antihypertensive medications included methyldopa, amlodipine and hydralazine. No patient received aspirin or metformin in this study.

Appointments were scheduled according to the routine. Maternal weight and blood pressure were assessed at every appointment and all mothers were screened for gestational diabetes according to the American Diabetes Association recommendations.

Obstetric and neonatal outcomes were obtained from the hospital records. Neonates were classified as small, appropriate or large for gestational age according to Olsen et al. growth curves.

Written informed consent was obtained from each participant after a full explanation of the study.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 2 consecutive pregnancy losses in the first trimester;
* losses should be documented by pathology or ultrasound-confirmed gestational sac.

Exclusion Criteria (any of the following):

* anatomic anomalies that may increase the risk of pregnancy losses, not amenable to surgical correction during pregnancy, such as uterine septum;
* antiphospholipid antibodies;
* prior second- or third-trimester losses;
* current multiple gestation;
* disabilities such as hemiplegia or paraplegia;
* renal or liver failure;
* conditions requiring a priori anticoagulation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 480 (Actual)
Dates: Start 2011-05; Primary Completion 2016-08 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Hoirisch-Clapauch, MD, PhD, Principal Investigator — Hospital Federal dos Servidores do Estado
Locations (1):
- Hospital Federal dos Servidores do Estado, Ministry of Health, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started on May 2011 and was stopped on April 2015.
Pre-assignment Details: Of 491 patients approached, 11 declined participation in the study and 480 were enrolled. Participants in the W+D arm were recommended lifestyle changes to be started when they wished to conceive. Only participants in both groups who managed to get pregnant were included in the study.
Groups:
- Walking & Dietary Modification (W&D): The intervention was standardized by training of research staff and should begin when participants wish to conceive. Careful instructions about walking speed and diet would be given to participants assigned to W&D at enrollment and at each consultation.
  Walking & dietary modification: 1. Daily walking at a moderate pace (4 km/h) > 40 min, 7/7. Those whose jobs required them to seat for long periods should walk 25-30 min twice a day, avoiding >12 h of physical inactivity. Walking may be replaced by stationary bicycle rides or swimming when convenient, such as near term.
  2. At least two daily servings of protein-rich food (≥ 4 g/kg of meat, poultry, fish or eggs) per day. Avoidance of high-carbohydrate, low-fiber meals, such as snacks, candies, fiber-free juices, coconut water, sugar-sweetened beverages or large amount of fruits. Sucralose could be used as a sweetener. Participants were recommended to use ondansetron for nausea and vomiting prevention
Period: Overall Study
Arm/Group | Walking & Dietary Modification (W&D) | Controls
Started | 178 | 171
Completed | 174 | 162
Not Completed | 4 | 9
Not completed — Multiple pregnancy | 2 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 0 | 4
Not completed — Lost the baby in a car accident | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Walking & Dietary Modification (W&D): The intervention was standardized by training of research staff and should begin when participants wish to conceive. Careful instructions about walking speed and diet would be given to participants assigned to W&D at enrolment and at each consultation.
  Walking & dietary modification: 1. Daily walking at a moderate pace (4 km/h) > 40 min, 7/7. Those whose jobs required them to seat for long periods should walk 25-30 min twice a day, avoiding >12 h of physical inactivity. Walking may be replaced by stationary bicycle rides or swimming when convenient, such as near term.
  2. At least two daily servings of protein-rich food (≥ 4 g/kg of meat, poultry, fish or eggs) per day. Avoidance of high-carbohydrate, low-fiber meals, such as snacks, candies, fiber-free juices, coconut water or sugar-sweetened beverages. Sucralose could be used as a sweetener. Participants were recommended to use ondansetron for nausea and vomiting prevention
- Total: Total of all reporting groups
Arm/Group | Walking & Dietary Modification (W&D) | Controls | Total
Number analyzed (Participants) | 174 | 162 | 336
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (7) | 30 (8) | 30 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 174 | 162 | 336
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 21 | 13 | 34
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 72 | 62 | 134
  White | 81 | 87 | 168
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 174 | 162 | 336
Normal or underweight (BMI <25 kg/m2) [Number; unit: participants] | 105 | 95 | 200
Owerweight (BMI 25-30 kg/m2) [Number; unit: participants] | 53 | 48 | 101
Obese (BMI > 30 kg/m2) [Number; unit: participants] | 16 | 19 | 35
Type 1 diabetes mellitus [Number; unit: participants] | 0 | 2 | 2
Chronic hypertension [Number; unit: participants] | 8 | 4 | 12
Women with live offspring [Number; unit: participants] | 36 | 28 | 64

OUTCOME MEASURES:

1. Primary Outcome: Take-home Baby Rate
Time Frame: End of pregnancy
Population: Since we excluded multiple gestations, there were 174 single pregnancies in group W&D and 162 in the control group.
Measure: Number; unit: babies
Groups:
- Walking & Dietary Modification (W&D): The intervention was standardized by training of research staff and should begin when participants wish to conceive. Careful instructions about walking speed and diet would be given to participants assigned to W&D at enrollment and at each consultation.
  Walking & dietary modification: 1. Daily walking at a moderate pace (4 km/h) > 40 min, 7/7. Those whose jobs required them to seat for long periods should walk 25-30 min twice a day, avoiding >12 h of physical inactivity. Walking may be replaced by stationary bicycle rides or swimming when convenient, such as near term.
  2. At least two daily servings of protein-rich food (≥ 4 g/kg of meat, poultry, fish or eggs) per day. Avoidance of high-carbohydrate, low-fiber meals, such as snacks, candies, fiber-free juices, coconut water, sugar-sweetened beverages and large amount of fruits. Sucralose could be used as a sweetener. Participants were recommended to use ondansetron for nausea and vomiting prevention
Arm/Group | Walking & Dietary Modification (W&D) | Controls
Number analyzed (Participants) | 174 | 162
babies | 152 | 83

2. Secondary Outcome: Gestational Diabetes Mellitus
Time Frame: Pregnancies reaching 24 weeks' gestation
Population: A total of 154 pregnancies in group W&D and 98 pregnancies in the control group reached 24 weeks of gestation.
Measure: Number; unit: mothers
Arm/Group | Walking & Dietary Modification (W&D) | Controls
Number analyzed (Participants) | 154 | 98
mothers | 4 | 17

3. Secondary Outcome: Preeclampsia
Time Frame: Pregnancies reaching 20 weeks' gestation
Population: A total of 154 pregnancies reached 20 weeks in group W&D and 98 in the control group.
Measure: Number; unit: mothers
Arm/Group | Walking & Dietary Modification (W&D) | Controls
Number analyzed (Participants) | 154 | 98
mothers | 8 | 22

4. Secondary Outcome: Mothers Who Used Heparin for Nephrotic Range Proteinuria or Placental Insufficiency
Time Frame: End of pregnancy
Measure: Number; unit: mothers
Arm/Group | Walking & Dietary Modification (W&D) | Controls
Number analyzed (Participants) | 174 | 162
mothers | 10 | 30

5. Secondary Outcome: Excessive Weight Gain
Description: Weight gain >13 kg for underweight, normal weight or overweight mothers and > 9 kg for obese mothers
Time Frame: End of term pregnancies
Population: A total of 148 pregnancies in group W&D and 57 pregnancies in the control group reached term.
Measure: Number; unit: mothers
Arm/Group | Walking & Dietary Modification (W&D) | Controls
Number analyzed (Participants) | 148 | 57
mothers | 12 | 21

6. Secondary Outcome: First-trimester Losses
Time Frame: 14 weeks of gestation
Population: Since we excluded multiple gestations, there were 174 single pregnancies in group W&D and 162 in the control group.
Measure: Number; unit: embryos
Arm/Group | Walking & Dietary Modification (W&D) | Controls
Number analyzed (Participants) | 174 | 162
embryos | 21 | 63

7. Secondary Outcome: Second and Third-trimester Losses
Time Frame: 28 weeks of gestation and end of gestation
Population: Since we excluded multiple gestations, there were 174 single pregnancies in group W&D and 162 in the control group.
Measure: Number; unit: fetuses
Arm/Group | Walking & Dietary Modification (W&D) | Controls
Number analyzed (Participants) | 174 | 162
fetuses | 0 | 7

8. Secondary Outcome: Live-born Children
Time Frame: End of pregnancy
Population: A total of 153 babies were born alive in group W&D and 91 in the control group.
Measure: Number; unit: babies
Arm/Group | Walking & Dietary Modification (W&D) | Controls
Number analyzed (Participants) | 174 | 162
babies | 153 | 91

9. Secondary Outcome: Babies Born at Term
Time Frame: End of pregnancy
Population: A total of 153 babies were born alive in group W&D and 91 in the control group.
Measure: Number; unit: babies
Arm/Group | Walking & Dietary Modification (W&D) | Controls
Number analyzed (Participants) | 153 | 91
babies | 138 | 57

10. Secondary Outcome: Appropriate-for-gestational Age Babies
Time Frame: End of pregnancy
Population: A total of 153 babies were born alive in group W&D and 91 in the control group.
Measure: Number; unit: babies
Arm/Group | Walking & Dietary Modification (W&D) | Controls
Number analyzed (Participants) | 153 | 91
babies | 141 | 56

11. Secondary Outcome: Neonates With Hypoglycemia
Description: Hypoglycemia was defined as any blood glucose concentration ≤ 40 mg/dL.
Time Frame: One, two and fours hours after birth
Population: A total of 153 babies were born alive in group W&D and 91 in the control group.
Measure: Number; unit: babies
Arm/Group | Walking & Dietary Modification (W&D) | Controls
Number analyzed (Participants) | 153 | 91
babies | 3 | 15

ADVERSE EVENTS:
Time Frame: Throughout pregnancy
Groups:
- Walking & Dietary Modification (W&D): The intervention was standardized by training of research staff and should begin when participants wish to conceive. Careful instructions about walking speed and diet will be given to participants assigned to W&D at enrollment and at each consultation.
  Walking & dietary modification: 1. Daily walking at a moderate pace (4 km/h) > 40 min, 7/7. Those whose jobs required them to seat for long periods should walk 25-30 min twice a day, avoiding >12 h of physical inactivity. Walking may be replaced by stationary bicycle rides or swimming when convenient, such as near term.
  2. At least two daily servings of protein-rich food (≥ 4 g/kg of meat, poultry, fish or eggs) per day. Avoidance of high-carbohydrate, low-fiber meals, such as snacks, candies, fiber-free juices, coconut water, sugar-sweetened beverages or large amount of fruits. Sucralose could be used as a sweetener. Participants were recommended to use ondansetron for nausea and vomiting prevention
Arm/Group | Walking & Dietary Modification (W&D) | Controls
All-Cause Mortality (participants affected / at risk) | 0/245 | 0/255
Serious Adverse Events (participants affected / at risk) | 0/245 | 0/255
Other Adverse Events (participants affected / at risk) | 1/245 | 0/255
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Walking & Dietary Modification (W&D) (N=245) | Controls (N=255)
Bone and joint injury (Musculoskeletal and connective tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
An important limitation of this study is that it did not assess the exact composition of the participants' diet.

Another limitation is that the use of heparin use was not controlled in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No